CLINICAL TRIAL: NCT04077541
Title: The Effects of a Nursing Trauma Care Bundle Combined With the Internet Platform in Patients With Extremity Injuries
Brief Title: the Effects of a Nursing Trauma Care Bundle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KMUHIRB-E(I)-20190203
Record Dates: First submitted 2019-08-26; First posted 2019-09-04 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Patient Portals
Keywords: trauma care bundles; internet platform; patients with extremity injuries; experimental design

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): The trauma care bundles combined with the internet platform.
  Interventions: Behavioral: internet platform
- The control group (No Intervention): Only trauma care bundles.

INTERVENTIONS:
Behavioral: internet platform — The trauma care bundles combined with the internet platform.
  Arms: The experimental group

SUMMARY:
To examine the effects of evidence-based care bundles combined with the internet platform in patients with extremity injuries. A longitudinal and two group experimental design will be used. Outcome measures for the trauma care bundles will use the Barthel's Index, the Posttraumatic Diagnostic Scale, and the World Health Organization Quality of Life questionnaire. The results may influence health policy and clinical practice, and a wide range of injured patient outcomes.

DETAILED DESCRIPTION:
Background: Over 50% of injuries are accompanied by musculoskeletal injuries that are life-threatening, require amputation or lead to major extremity dysfunctions. Some barriers exist to deliver evidence-based care in the trauma group. Based on recent research findings, this project will be an evidence-based project and evaluation of care bundles combined with e health care to establish and refine evidence-based care guidelines for patients with extremity injuries in Taiwan.

Aims: To examine the effects of evidence-based care bundles combined with the internet platform in patients with extremity injuries.

Methods: A longitudinal and two group experimental design will be used. The trauma care bundles combined with internet platform will be implemented over 24-hour admission and ended in 10-14 days after hospital discharge. Participants will be patients with extremity injuries that meet the criteria. The experimental group and the control group will be given the same routine care except for the trauma care bundles. Both groups will be followed up at 3 and 6 months after hospital discharge. Fifty-eight participants for each group will be expected. The generalized estimating equations will be used to analyze the data. Outcome measures for the trauma care bundles will use the Barthel's Index, the Posttraumatic Diagnostic Scale, and the World Health Organization Quality of Life questionnaire.

Expected outcomes: This is an innovation project as it combines a comprehensive trauma care bundles with internet platform, and applied in the biggest injury population in Taiwan. It may be the pioneer study to integrate care bundle and e-health care in trauma care. The results may influence health policy and clinical practice, and a wide range of injured patient outcomes. The internet platform established by the research team may be an important template for domestic e-health in hospital-based settings and long-term care facilities.

ELIGIBILITY:
Inclusion Criteria:

* ISS (Injury Severe Score)>9
* Agree to participate in this examination for 6 months after discharge
* Accidental extremity injuries
* Have a smart phone and access to the Internet

Exclusion Criteria:

* Discharged within 24 hours
* Cognitive dysfunction and unable to provide formal consent
* Severe brain damage
* Burned patient
* Severe psychosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
the Numeric Pain Rating Scale | at 1 day before hospital discharge
  The NPRS is a one-dimensional measure of pain intensity in adults. A NPRS has similar anchors at the extremes but offers numbers from 0 through 10. It is well known and broadly used scale in clinical settings. It also used to be applied in post injury pain
the Numeric Pain Rating Scale | at 10 to 14 days after hospital discharge
  The NPRS is a one-dimensional measure of pain intensity in adults. A NPRS has similar anchors at the extremes but offers numbers from 0 through 10. It is well known and broadly used scale in clinical settings. It also used to be applied in post injury pain
the Barthel's Index | at 1 day before hospital discharge
  The BI will be used to measure functional disabilities patients with extremity injury. The BI, organically developed by Mahoney and Barthel (1965), assesses BADL in terms of respondent abilities related to feeding, bathing, grooming, dressing, bowel and bladder control, toilet use, transfer, mobility, and stair use. The BI has 30 items with scores range from 0 to 100, with higher scores representing higher independence in performing BADLs. A total BI score of 0 to 20 correlates with total dependence, 21 to 60 correlates with severe dependence, 61 to 90 correlates with moderate dependence, 91 to 99 correlates with slight dependence, and 100 correlates with total independence. The Chinese version was applied in older populations, with Cronbach's alpha ranging from 0.79 to .085 (Shyu, Tang, Tsai, Liang, & Chen, 2006). The Cronbach's alpha for this current project will be retested using the injury group.
the Barthel's Index | at 10 to 14 days after hospital discharge
  The BI will be used to measure functional disabilities patients with extremity injury. The BI, organically developed by Mahoney and Barthel (1965), assesses BADL in terms of respondent abilities related to feeding, bathing, grooming, dressing, bowel and bladder control, toilet use, transfer, mobility, and stair use. The BI has 30 items with scores range from 0 to 100, with higher scores representing higher independence in performing BADLs. A total BI score of 0 to 20 correlates with total dependence, 21 to 60 correlates with severe dependence, 61 to 90 correlates with moderate dependence, 91 to 99 correlates with slight dependence, and 100 correlates with total independence. The Chinese version was applied in older populations, with Cronbach's alpha ranging from 0.79 to .085 (Shyu, Tang, Tsai, Liang, & Chen, 2006). The Cronbach's alpha for this current project will be retested using the injury group.
the Barthel's Index | at 3 months after hospital discharge
  The BI will be used to measure functional disabilities patients with extremity injury. The BI, organically developed by Mahoney and Barthel (1965), assesses BADL in terms of respondent abilities related to feeding, bathing, grooming, dressing, bowel and bladder control, toilet use, transfer, mobility, and stair use. The BI has 30 items with scores range from 0 to 100, with higher scores representing higher independence in performing BADLs. A total BI score of 0 to 20 correlates with total dependence, 21 to 60 correlates with severe dependence, 61 to 90 correlates with moderate dependence, 91 to 99 correlates with slight dependence, and 100 correlates with total independence. The Chinese version was applied in older populations, with Cronbach's alpha ranging from 0.79 to .085 (Shyu, Tang, Tsai, Liang, & Chen, 2006). The Cronbach's alpha for this current project will be retested using the injury group.
the Barthel's Index | at 6 months after hospital discharge
  The BI will be used to measure functional disabilities patients with extremity injury. The BI, organically developed by Mahoney and Barthel (1965), assesses BADL in terms of respondent abilities related to feeding, bathing, grooming, dressing, bowel and bladder control, toilet use, transfer, mobility, and stair use. The BI has 30 items with scores range from 0 to 100, with higher scores representing higher independence in performing BADLs. A total BI score of 0 to 20 correlates with total dependence, 21 to 60 correlates with severe dependence, 61 to 90 correlates with moderate dependence, 91 to 99 correlates with slight dependence, and 100 correlates with total independence. The Chinese version was applied in older populations, with Cronbach's alpha ranging from 0.79 to .085 (Shyu, Tang, Tsai, Liang, & Chen, 2006). The Cronbach's alpha for this current project will be retested using the injury group.
the Posttraumatic Diagnostic Scale | at 3 months after hospital discharge
  The PTDS is a self-report instrument for post traumatic syndrome that is simple to administer and has demonstrated good psychometric properties. The PTSD will not use to diagnose if injured patients have psychological illnesses. It will be applied in measuring how and what post traumatic symptoms that patients will have after injuries. The scale is a structured interview for assessing PTSD diagnostic status and symptom. The degree of severity is rated on a five-point scale scoring with zero: not at all, one: once per week or less / a little, two: 2 to 3 times per week / somewhat, three: 4 to 5 times per week / a lot, and four: 6 or more times a week / severe (Pynoos et al., 1993). This instrument was not only broadly used in patients with mental illnesses, but also used in patients with vehicle accidents domestically (Wang, 2013). The Cronbach's alpha for the current study will be retested using the injury group.
the Posttraumatic Diagnostic Scale | at 6 months after hospital discharge
  The PTDS is a self-report instrument for post traumatic syndrome that is simple to administer and has demonstrated good psychometric properties. The PTSD will not use to diagnose if injured patients have psychological illnesses. It will be applied in measuring how and what post traumatic symptoms that patients will have after injuries. The scale is a structured interview for assessing PTSD diagnostic status and symptom. The degree of severity is rated on a five-point scale scoring with zero: not at all, one: once per week or less / a little, two: 2 to 3 times per week / somewhat, three: 4 to 5 times per week / a lot, and four: 6 or more times a week / severe (Pynoos et al., 1993). This instrument was not only broadly used in patients with mental illnesses, but also used in patients with vehicle accidents domestically (Wang, 2013). The Cronbach's alpha for the current study will be retested using the injury group.
the WHOQOL-BREF | at 3 months after hospital discharge
  The World Health Organization Quality of Life questionnaire (WHOQOL-BREF) will be used to measure HRQOL. Six popular generic instruments of HRQOL are commonly used as disability outcome measures, some of them were developed later were tested trans-culturally in extensive research programs such as the WHOQOL-BREF (Yao, 2000). The WHOQOL-BREF is a 28-tem scale that is measure along with 4 domains including physical, psychological, social relationship and environment. Scores range from 1 to 5 with higher scores indicating higher quality of life (The WHOQOL Taiwan Group, 2000). The reliability and validity of the Chinese WHOQOL-BREF have been tested in various clinical settings.
the WHOQOL-BREF | at 6 months after hospital discharge
  The World Health Organization Quality of Life questionnaire (WHOQOL-BREF) will be used to measure HRQOL. Six popular generic instruments of HRQOL are commonly used as disability outcome measures, some of them were developed later were tested trans-culturally in extensive research programs such as the WHOQOL-BREF (Yao, 2000). The WHOQOL-BREF is a 28-tem scale that is measure along with 4 domains including physical, psychological, social relationship and environment. Scores range from 1 to 5 with higher scores indicating higher quality of life (The WHOQOL Taiwan Group, 2000). The reliability and validity of the Chinese WHOQOL-BREF have been tested in various clinical settings.

CONTACTS AND LOCATIONS:
Overall Officials: Bih-O Lee, PHD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan